CLINICAL TRIAL: NCT02008435
Title: Increasing the Effectiveness of the Diabetes Prevention Program Through If-then Plans and Mental Practice: A Parallel Randomized Trial
Brief Title: Increasing the Effectiveness of the Diabetes Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Barbel Knauper, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MOP-123242
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Overweight; Obesity
Keywords: Group-delivered Diabetes Prevention Program; Obesity; Overweight; Lifestyle change; Healthy eating; Weight loss; Exercise; Cognitive-behavioral intervention; Implementation intentions; Mental imagery; Mental practice; If-then plans
MeSH Terms: conditions — Overweight; Obesity; Weight Loss; Motor Activity | interventions — Weight Reduction Programs

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enriched GLB (Experimental): This arm aims to increase the effectiveness of the Group Lifestyle Balance (GLB) program by integrating habit formation techniques, namely if-then plans and their mental practice, into the program.
  Interventions: Behavioral: Enriched GLB
- Standard GLB (Active Comparator): This arm is the standard Group Lifestyle Balance (GLB) program, which is the group version of the Diabetes Prevention Program developed by the NIH.
  Interventions: Behavioral: Standard GLB

INTERVENTIONS:
Behavioral: Enriched GLB — Habit formation techniques, namely if-then plans and their mental practice are being added to the standard Group Lifestyle Balance program.
  Other Names: Diabetes Prevention Program; weight loss program; implementation intentions; mental imagery
  Arms: Enriched GLB
Behavioral: Standard GLB — This arm is the standard Group Lifestyle Balance program
  Other Names: Diabetes Prevention Program; weight loss program
  Arms: Standard GLB

SUMMARY:
The Diabetes Prevention Program (DPP) is highly effective in promoting weight loss in overweight and obese individuals (e.g., 7% average loss of body weight), and thereby reducing the risk of developing weight-related health consequences. One-on-one DPP sessions, however, are costly and the group-delivered DPP version, the Group Lifestyle Balance program (GLB), is less effective (4% average loss of body weight). The aim of this two-arm parallel randomized controlled trial is to increase the effectiveness of the GLB by integrating habit formation techniques, namely if-then plans and their mental practice, into the program. The study will provide evidence-based data on the effectiveness of an enhanced GLB intervention in promoting weight loss and in reducing weight-related risk factors for chronic health problems.

DETAILED DESCRIPTION:
Please see brief summary.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* ages of 18 and 75
* overweight or obese (BMI 28-45 kg/m2)
* sedentary (< 200 min/week of moderate or vigorous exercise)
* waist circumference of >= 88cm for women and >= 102cm for men

Exclusion Criteria:

* diabetes (hemoglobin A1c < 7.0%).
* taking the medication metformin (used for treating pre-diabetes or diabetes)
* having been pregnant in the past 6 months or planning on becoming pregnant in the next 2 years
* currently undergoing treatment for cancer
* using medication that affects body weight (e.g., loop diuretics)
* being unable to participate in regular moderate physical activity
* having severe uncontrolled hypertension (> 190/100mm Hg)
* being unable to communicate in English or French
* being diagnosed with bulimia nervosa, currently active major depression, or other severe psychiatric disease (including dementia);
* suffering from a heart attack, stroke, or heart failure within the past 6 months
* experiencing excessive weight loss (more than 10 pounds or 4.54 kilograms) in the past 3 months
* currently participating in another weight loss program
* having had bariatric surgery in the past 2 years or plans on getting it in the near future
* planning on moving away from Montreal within the next year
* having another member of one's household enrolled in the program.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Percent body weight loss | 3 months after beginning of the intervention
  The primary outcome will be percent body weight loss from baseline to 3 months after the beginning of the intervention. Weight in kg.

SECONDARY OUTCOMES:
Percent body weight loss | 12 months
  Percent body weight loss 12 months after the beginning of the intervention. Weight in kg.
Percent body weight loss | 24 months
  Percent body weight loss 24 months after the beginning of the intervention. Weight in kg.
Personal weight loss goal | 3 months
  Reaching percent body weight loss goal (7% of body weight) from baseline to 3 months after the beginning of the intervention. Weight in kg.
Personal weight loss goal | 12 months
  Reaching percent body weight loss goal (7% of body weight) 12 months after the beginning of the intervention. Weight in kg.
Personal weight loss goal | 24 months
  Reaching percent body weight loss goal (7% of body weight) 24 months after the beginning of the intervention. Weight in kg.
Personal exercise goal | 3 months
  Reaching exercise goal (150 min/week) from baseline to 3 months after the beginning of the intervention. Sum of minutes over 7 days.
Personal exercise goal | 12 months
  Reaching exercise goal (150 min/week) 12 months after the beginning of the intervention. Sum of minutes over 7 days.
Personal exercise goal | 24 months
  Reaching exercise goal (150 min/week) 24 months after the beginning of the intervention. Sum of minutes over 7 days.
Waist circumference | 3 months
  Risk factor for chronic health problems.
Waist circumference | 12 months
  Risk factor for chronic health problems.
Waist circumference | 24 months
  Risk factor for chronic health problems.
Hemoglobin A1c levels | 3 months
  Risk factor for chronic health problems.
Hemoglobin A1c levels | 12 months
  Risk factor for chronic health problems.
Hemoglobin A1c levels | 24 months
  Risk factor for chronic health problems.
Blood pressure | 3 months
  Risk factor for chronic health problems.
Blood pressure | 12 months
  Risk factor for chronic health problems.
Blood pressure | 24 months
  Risk factor for chronic health problems.
Total cholesterol/HDL ratio | 3 months
  Risk factor for chronic health problems.
Total cholesterol/HDL ratio | 12 months
  Risk factor for chronic health problems.
Total cholesterol/HDL ratio | 24 months
  Risk factor for chronic health problems.
Physical activity duration | 3 months
  Total minutes per week.
Physical activity duration | 12 months
  Total minutes per week.
Physical activity duration | 24 months
  Total minutes per week.
Number of steps taken per week | 3 months
  Steps taken per week, recorded using a pedometer.
Number of steps taken per week | 12 months
  Steps taken per week, recorded using a pedometer.
Number of steps taken per week | 24 months
  Steps taken per week, recorded using a pedometer.
Exercise stress test (EST) | 3 months

OTHER OUTCOMES:
Self-Report Index of Habit Strength | 3 months
  Self-monitoring and behaviors
Self-Report Index of Habit Strength | 12 months
  Self-monitoring and behaviors
Self-Report Index of Habit Strength | 24 months
  Self-monitoring and behaviors
Habit formation indices of weight tracking | 3 months
  Frequency of weight tracking.
Habit formation indices of weight tracking | 12 months
  Frequency of weight tracking.
Habit formation indices of weight tracking | 24 months
  Frequency of weight tracking.
Habit formation indices of physical activity tracking | 3 months
  Frequency of physical activity tracking.
Habit formation indices of physical activity tracking | 12 months
  Frequency of physical activity tracking.
Habit formation indices of physical activity tracking | 24 months
  Frequency of physical activity tracking.
Habit formation indices of fat grams and calorie tracking | 3 months
  Frequency of food tracking.
Habit formation indices of fat grams and calorie tracking | 12 months
  Frequency of food tracking.
Habit formation indices of fat grams and calorie tracking | 24 months
  Frequency of food tracking.

CONTACTS AND LOCATIONS:
Overall Officials: Barbel Knauper, PhD, Principal Investigator — McGill University; Ilka Lowensteyn, PhD, Study Director — McGill University; Lawrence Joseph, PhD, Study Director — McGill University; Aleksandra Luszczynska, PhD, Study Director — University of Colorado, Denver; Steven Grover, MD, Study Director — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Knauper B, Shireen H, Carriere K, Frayn M, Ivanova E, Xu Z, Lowensteyn I, Sadikaj G, Luszczynska A, Grover S; McGill CHIP Healthy Weight Program Investigators. The effects of if-then plans on weight loss: results of the 24-month follow-up of the McGill CHIP Healthy Weight Program randomized controlled trial. Trials. 2020 Jan 7;21(1):40. doi: 10.1186/s13063-019-4014-z. PMID 31910891
- [Derived] Knauper B, Carriere K, Frayn M, Ivanova E, Xu Z, Ames-Bull A, Islam F, Lowensteyn I, Sadikaj G, Luszczynska A, Grover S; McGill CHIP Healthy Weight Program Investigators. The Effects of If-Then Plans on Weight Loss: Results of the McGill CHIP Healthy Weight Program Randomized Controlled Trial. Obesity (Silver Spring). 2018 Aug;26(8):1285-1295. doi: 10.1002/oby.22226. Epub 2018 Jun 28. PMID 29956503
- [Derived] Knauper B, Ivanova E, Xu Z, Chamandy M, Lowensteyn I, Joseph L, Luszczynska A, Grover S. Increasing the effectiveness of the Diabetes Prevention Program through if-then plans: study protocol for the randomized controlled trial of the McGill CHIP Healthy Weight Program. BMC Public Health. 2014 May 18;14:470. doi: 10.1186/1471-2458-14-470. PMID 24885388